CLINICAL TRIAL: NCT05322668
Title: Evaluation of the Tolerance of Cyto-selective Difluoroethane-based Cryotherapy
Brief Title: Tolerance of Cyto-selective Difluoroethane-based Cryotherapy
Acronym: AGILE3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Collaborators: INNOVSOLUTION (Unknown); CEISO (Industry); Dermatech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (CS4_3)IVYTOP-N°21D588A0003
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-03

CONDITIONS: Solar Lentigo
Keywords: Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Condition 1 (Experimental): All the subjects will receive all the treatment in the same order.
  The following prototypes will be applied on hands areas:
  Application of the prototype (812A-v1) at Day 0, Application of the prototype (812C-v1) at Day 0, Application of the prototype (812D-v1) at Day 0, Application of the prototype (812F-v1) at Day 0,
  Interventions: Device: Prototypes (812A-v1), (812C-v1), (812D-v1) and (812F-v1)

INTERVENTIONS:
Device: Prototypes (812A-v1), (812C-v1), (812D-v1) and (812F-v1) — All the subjects will receive all the treatment in the same order.
  On each hand 2 devices will be attributed as follow:
  * Prototypes (812A-v1) will be applied on an area of the back of the patient's right hand, on healthy skin
  * Prototypes (812C-v1) will be applied on an area of the back of the patient's right hand, on healthy skin
  * Prototypes (812D-v1) will be applied on an area of the back of the patient's left hand, on healthy skin
  * Prototypes (812F-v1) will be applied on an area of the back of the patient's left hand, on healthy skin

SUMMARY:
Cryotherapy is more and more used to improve skin appearance. Devices using difluoroethane, manufactured by CRYONOVE PHARMA, are already available on the local and international markets, e.g. CRYOBEAUTY MAINS and CRYOBEAUTY CORPS.

However, the cryogenic gas (conventional cryotherapy - liquid nitrogen) creates a dermabrasion of the skin surface and person receiving this kind of treatment presents an impaired skin during a few days following the treatment as temporary damage of stratum corneum, erythema, scars, burns.

Following the side effects occurring after conventional cryotherapy application, it seems interesting for the sponsor to select other sequences of a cryogenic spray (4 prototypes of devices) which could be used for lentigo treatment with a same benefit for the consumers without any safety outcomes.

This study will assess the use of different prototypes with a sequence of application of cryogenic gas which reaches a higher temperature than those which used with the reference device, in order to increase the acceptability of the device.

(CS4_3) proof of concept, interventional, monocentric, aims to evaluate the tolerance of cryotherapy treatments applied on healthy skin on the back of the hands.

The main objective of the study is to evaluate on phototype V and VI, the tolerance of 4 different conditions of cryotherapy treatments (4 prototypes) applied on healthy skin on the back of the hands.

DETAILED DESCRIPTION:
Prototypes (812A-v1), (812C-v1), (812D-v1) and (812F-v1) will be applied on hands areas by the same order for all volunteers using a reposition mask. On each hand 2 devices will be attributed starting from the middle point of the hand toward to the lateral internal and lateral external edges of the hand. The distance between 2 treatment areas will be 2 cm.

Each area will be treated 1 time during the study at D0. The treatment will starts from right hand with prototypes (812A-v1) and (812C-v1), then left hands with the prototypes (812D-v1) and (812F-v1) .

Prior to any study device application, the dermatologist will assess the adverse events.

The dermatologist will verify that the skin has not been treated by cosmetic products (no presence of cream that could interfere with the treatment) and is dry.

The procedure will take place at the investigation site. An operator previously trained by the dermatologist will apply the study device to the patient's hand.

Subjects will lie down and the device will be administered upside down.

The prototypes will be applied 10 minutes apart so that pain can be measured without interference from application to application.

ELIGIBILITY:
Inclusion Criteria:

* Female or male.
* Ages > 18.
* Phototype V et VI (according with Fitzpatrick scale)
* Agreeing not to be exposed to the sun (or artificial UV) during the study.
* Informed, having undergone a general clinical examination attesting to his/her ability to participate in the study.
* Having given written consent for participation in the study.
* No suspicion of carcinoma after investigation by a dermatologist.

Exclusion Criteria:

* Having performed cosmetic treatments (exfoliants, scrubs or self-tanners, facials, UV ...) in the month before the start of the study, at the level of the hand.
* Having applied a depraving product in the month prior to the start of the study, at the hands (except cleansing products).
* Having performed cosmetic treatments in a dermatologist (laser, IPL (Intensed pulsed light), peeling, creams, cryotherapy ...), on the hands in the last 6 months.
* With dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (people with diabetes or circulatory problems,allergic to cold, Raynaud's syndrome...).
* Receiving treatment by general or local (dermo corticoids, corticosteroids, diuretics ...) likely to interfere with the evaluation of the parameter studied.
* Participating in another study or being excluded from a previous study.
* Unable to follow the requirements of the protocol.
* Vulnerable: whose ability or freedom to give or refuse consent is limited.
* Major protected by law (tutorship, curatorship, safeguarding justice...).
* People unable to understand, read and write English/French/Ukrainian language. However, the impartial witness will be introduced to current study to make translations if necessary, during all course of the study for each volunteer and respective section for signature and date will be implemented to the "Information Sheet and Informed Consent Form".
* Unable to be contacted urgently over the phone.

For female subjects:

* Pregnant woman (or wishing to be pregnant during study) or while breastfeeding.
* A woman, who does not use effective methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline skin hyperpigmentation | Day 0, Day 2, Day 7, Day 21, Day 56
  This outcome is a tolerance assessment criteria. Clinical evaluation of hyperpigmentation on each selected and treated area will be performed by a Dermatologist using the Investigator's Global Assessment likert 6 points scale ranged from 0 to 5: 0=Clear of hyperpigmentation, 1= Almost clear of hyperpigmentation, 2=mild, but noticeable hyperpigmentation, 3=moderate hyperpigmentation (medium brown in quality), 4=severe hyperpigmentation (dark brown in quality), 5= very severe hyperpigmentation (very dark brown, almost black in quality)
Change from baseline skin hypopigmentation | Day 0, Day 2, Day 7, Day 21, Day 56
  This outcome is a tolerance assessment criteria. Clinical evaluation of hypopigmentation on each selected and treated area will be performed by a Dermatologist using a likert 5 points scale ranged from 0 to 4: 0=no hypopigmented lesion, 1= very slight area of hypopigmentation of very small size and very slightly fairer than the surrounding skin, 2= slight area of hypopigmentation of small size and slightly fairer than the surrounding skin, 3= moderate : area of hypopigmentation of moderate size and much fairer than the surrounding skin, 4= severe : area of hypopigmentation of large size and much fairer than the surrounding skin.
Change from baseline skin appearance (Edemas, blisters, bubbles, scars, erythema) | Day 0, Day 2, Day 7, Day 21, Day 56
  his outcome is a tolerance assessment criteria. Clinical visual evaluation of selected area and surrounded spotless skin area around the spot skin will be performed. A likert scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Change from baseline skin sensation (itching, tingling, burning sensations) | Day 0, Day 2, Day 7, Day 21, Day 56
  This outcome is a tolerance assessment criteria. Clinical visual evaluation of selected lentigo spots and around the spot skin will be performed. A likert scale in 5 points (0 to 4) will be used : 0=none; 1=very mild; 2=mild; 3=moderate; 4=severe.
Post treatment pain | Day 0
  This outcome is a tolerance assessment criteria. The pain of the treatment will be assessed by the VAS (Visual Analogue Scale). Pain intensity is measured in millimeters by the distance from the position of the mark to the "no pain" extremity.
Other unexpected events | at Day0, Day2, Day7, Day21 and Day56
  This outcome concerns the occurence of the adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- VIDNOVLENNYA medical center, Zhytomyr, Ukraine